CLINICAL TRIAL: NCT03694431
Title: A Non-Inferiority Comparative Effectiveness Trial of Home-Based Palliative Care in Older Adults
Brief Title: Comparative Trial of Home-Based Palliative Care
Acronym: HomePal
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low intervention uptake, lack of substitution of video for home visits, and study sites' decision to expand telehealth use in response to payment changes
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PLC-1609-36108
Record Dates: First submitted 2018-09-27; First posted 2018-10-03 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Cancer; Chronic Obstructive Pulmonary Disease; Heart Failure; Dementia; End Stage Liver Disease; End Stage Renal Disease; Neuromuscular Diseases
MeSH Terms: conditions — Neoplasms; Pulmonary Disease, Chronic Obstructive; Heart Failure; Dementia; End Stage Liver Disease; Kidney Failure, Chronic; Neuromuscular Diseases

STUDY DESIGN:
Intervention Model Description: Randomization of registered nurses stratified by site (n=15) to either standard or tech-supported HBPC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard HBPC (Active Comparator): Patients and caregivers in standard HBPC will continue to receive usual care from the palliative care team which includes home visits
  Interventions: Other: Standard HBPC
- Tech-supported HBPC (Experimental): Patients and caregivers in tech-supported HBPC will receive synchronous video visits with a provider (physician or nurse practitioner) while the nurse is in the patient's home. Home visits by the palliative care team will be determined based on patients/caregivers' needs.
  Interventions: Other: Tech-supported HBPC

INTERVENTIONS:
Other: Tech-supported HBPC — Palliative care provided consistent with recommendations from the National Consensus Project for Quality Palliative Care
  Arms: Tech-supported HBPC
Other: Standard HBPC — Palliative care provided consistent with recommendations from the National Consensus Project for Quality Palliative Care
  Arms: Standard HBPC

SUMMARY:
Background: To effectively alleviate suffering and improve quality of life for patients with serious illness and their caregivers, palliative care (PC) services must be offered across multiple settings. Research is needed to determine how best to optimize home-based palliative care (HBPC) services to meet the needs of individuals with high symptom burden and functional limitations.

Aim: The investigators will compare a standard HBPC model that includes routine home visits by a nurse and provider with a more efficient tech-supported HBPC model that promotes timely inter-professional team coordination via synchronous video consultation with the provider while the nurse is in the patient's home. The investigators hypothesize that tech-supported HBPC will be as effective as standard HBPC.

Design: Cluster randomized trial. Registered nurses (n~130) will be randomly assigned to the tech-supported or standard HBPC model so that half of the patient-caregiver dyads will receive one of the two models.

Setting/Participants: Kaiser Permanente (15 Southern California and Oregon sites). Patients (n=10,000) with any serious illness and a prognosis of 1-2 years and their caregivers (n=4,800)

Methods: Patients and caregivers will receive standard PC services: comprehensive needs assessment and care planning, pain and symptom management, education/skills training, medication management, emotional/spiritual support; care coordination, referral to other services, and 24/7 phone assistance.

Results: Primary patient outcomes: symptom improvement at 1 month and days spent at home in the last six months of life; caregiver outcome: perception of preparedness for caregiving.

Conclusion: Should the more efficient tech-supported HBPC model achieves comparable improvements in outcomes that matter most to patients and caregivers, this would have a lasting impact on PC practice and policy.

ELIGIBILITY:
Patient Inclusion Criteria:

* Serious illness with 12-24 month life expectancy
* Homebound
* Need for skilled nursing care (only at KP Southern California)
* English or Spanish speakers

Patient Exclusion Criteria:

- Currently receiving HBPC

Caregiver Inclusion Criteria:

* Non-professional family, friend or other caregiver
* English or Spanish speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3999 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Symptom severity (total score) using the Edmonton Symptom Assessment Scale (ESAS) | Change from baseline to 1 month
  The ESAS is a 10-item survey measuring symptom severity. Scores range from 0-100 with higher scores indicating worse symptoms.
Days at home in the last 180 days of life among patients surviving at least 180 days after enrolling in HBPC | Baseline to 12 months
Caregiver preparedness for caregiving using the Preparedness for Caregiving Scale | Change from baseline to 1 month
  The Preparedness for Caregiving Scale is a 9-item survey measuring caregivers' perception of their preparedness for caregiving. Scores range from 0-36 with higher scores indicating higher perception of preparedness

SECONDARY OUTCOMES:
Days at home between study enrollment and death or study completion (365 days) | Variable, up to 12 months
Patient quality of life measured with the PROMIS-10 survey | Change from baseline to 1 and 6 months
  The PROMIS-10 is a 10-item survey measuring general health related quality of life. Scores range from 0-100 with higher scores indicating better quality of life
Patient general distress measured with the distress thermometer | Change from baseline to 1 and 6 months
  Scores for this single item distress thermometer range from 0-10 with higher scores indicating greater distress
Palliative performance scale will be measured using all data available from routine clinical practice as documented in the electronic medical record (EMR) | Baseline and variable time periods due to reliance on available data from the EMR
  The Palliative Performance Scale measures overall functional status. A clinician completes this assessment using a scale of 0-100 with higher scores indicating better functional performance
Patient satisfaction-care experience measured by a study-specific survey | 1 and 6 months
  This 8-item satisfaction-care experience survey was developed specifically to measure satisfaction and care experience with home-based palliative care.
Patient acute and post-acute care utilization | Baseline to 12 months
  Frequency of hospitalizations, emergency department visits and skilled nursing facility stay
Patient outpatient health care utilization | Baseline to 12 months
  Frequency of primary and specialty care visits
Patient enrollment in and days on hospice before death | Baseline to 12 months
Patient death | Baseline to 12 months
Caregiver quality of life measured with the PROMIS-10 | Change from baseline to 1 and 6 months
  The PROMIS-10 is a 10-item survey measuring general health related quality of life. Scores range from 0-100 with higher scores indicating better quality of life
Caregiver burden measured with the Zarit-12 Caregiver Burden Scale | Change from baseline to 1 and 6 months
  The Zarit-12 is a 12-item survey measuring caregiver burden. Scores range from 0-48 with higher scores indicating greater caregiver burden
Caregiver acute and post-acute care utilization | Baseline to 12 months
  Frequency of hospitalizations, emergency department visits and skilled nursing facility stay for caregivers who are members of Kaiser Permanente
Caregiver outpatient health care utilization | Baseline to 12 months
  Frequency of primary and specialty care visits for caregivers who are members of Kaiser Permanente
HBPC clinician perception of facilitators and barriers to implementation of HBPC services | Yearly, up to four years
  Study specific survey (under development)

CONTACTS AND LOCATIONS:
Overall Officials: Huong Q Nguyen, PhD, Principal Investigator — Kaiser Permanente; Richard A Mularski, MD, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - Kaiser Permanente Southern California, Pasadena, California
  - Kaiser Permanente Northwest, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen HQ, Haupt EC, Duan L, Hou AC, Wang SE, Mariano JD, Lee JA, McMullen C. Hospital utilisation in home palliative care: caregiver health, preparedness and burden associations. BMJ Support Palliat Care. 2022 Jan 25:bmjspcare-2021-003455. doi: 10.1136/bmjspcare-2021-003455. Online ahead of print. PMID 35078873
- [Derived] Mularski RA, Mittman B, Haupt E, Wang S, Scholle S, McMullen C, Henry M, Shen E, Nguyen HQ; HomePal Research Group. Performance of Patient-Reported Outcome Measures in a Large Pragmatic Trial of Home-Based Palliative Care (HomePal): Methodological and Practical Considerations for Embedded Patient-Centered Design. J Palliat Med. 2022 Apr;25(4):620-627. doi: 10.1089/jpm.2021.0164. Epub 2021 Nov 3. PMID 34735285
- [Derived] Nguyen HQ, Mularski RA, Edwards PE, Lynn J, Machado MT, McBurnie MA, McMullen C, Mittman BS, Reinke LR, Shen E, Wang SE, Werch HS; HomePal Research Group. Protocol for a Noninferiority Comparative Effectiveness Trial of Home-Based Palliative Care (HomePal). J Palliat Med. 2019 Sep;22(S1):20-33. doi: 10.1089/jpm.2019.0116. PMID 31486724